CLINICAL TRIAL: NCT02275507
Title: Non-Invasive Hemoglobin Monitoring of Women Undergoing Cesarean Delivery
Status: Completed | Type: Observational
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Joseph Chappelle, Assistant Professor, Stony Brook University
Other Study IDs: 613231
Record Dates: First submitted 2014-10-23; First posted 2014-10-27 (Estimated); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Complications of Pregnancy, Childbirth and the Puerperium
MeSH Terms: conditions — Pregnancy Complications

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Women Undergoing Scheduled Cesarean Delivery: We will be recruiting women who are scheduled for an elective repeat or primary cesarean delivery.
  Interventions: Device: Masimo Rainbow Sensor

INTERVENTIONS:
Device: Masimo Rainbow Sensor — Non-Invasive Hemoglobin Measurement

SUMMARY:
The purpose of this study is to determine the normal hemoglobin curve during cesarean delivery and for the first 24 hours after surgery to aid in the creation of an algorithm to detect life-threatening bleeding earlier.

DETAILED DESCRIPTION:
Acute and life threatening blood loss is the most common cause of morbidity and mortality for pregnancy women in the US. To date, the only means we have of monitoring the amount of blood loss during a delivery is by the physician estimating the amount. This has been shown to not be very accurate and leads to confusion on when and how much a women should be transfused during a hemorrhage. New devices have been developed over the last few years to monitor blood levels in a accurate and non-invasive fashion. We aim here to use a non-invasive blood monitoring system to evaluate normal blood loss in women undergoing scheduled cesarean delivery. We hope that this will allow us to create a baseline that can be used in subsequent studies to identify women who are losing more blood than normal so that we may intervene faster and avoid unnecessary morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing scheduled cesarean delivery

Exclusion Criteria:

* Blood disorders (i.e. thalassemia, sickle cell), hypertensive disorders, obstetric risk factors for hemorrhage

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: women who are scheduled for an elective repeat or primary cesarean delivery. We will exclude women at high-risk for hemorrhage, thalassemia major, sickle cell disease, or women with hypertensive disorders
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2014-10-15 (Actual); Primary Completion 2016-10-30 (Actual); Study Completion 2016-10-30 (Actual)

PRIMARY OUTCOMES:
Decrease in Hemoglobin over time | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Chappelle, MD, Principal Investigator — Stony Brook University Hospital
Locations (1):
- Stony Brook University Hospital, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chamos C, Vele L, Hamilton M, Cecconi M. Less invasive methods of advanced hemodynamic monitoring: principles, devices, and their role in the perioperative hemodynamic optimization. Perioper Med (Lond). 2013 Sep 17;2(1):19. doi: 10.1186/2047-0525-2-19. PMID 24472443
- [Background] Butwick A, Hilton G, Carvalho B. Non-invasive haemoglobin measurement in patients undergoing elective Caesarean section. Br J Anaesth. 2012 Feb;108(2):271-7. doi: 10.1093/bja/aer373. Epub 2011 Nov 23. PMID 22116296